CLINICAL TRIAL: NCT05985863
Title: Clinical Research of Human Umbilical Cord Mesenchymal Stem Cell Transplantation for The Treatment of Acute-on-Chronic Liver Failure
Brief Title: Human Umbilical Cord Mesenchymal Stem Cell Transplantation for The Treatment of Acute-on-Chronic Liver Failure
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing 302 Hospital (Other)
Collaborators: Shulan (Hang Zhou) Hospital (Unknown); BeijingYouan Hospital (Unknown); Shenzhen Third People's Hospital (Other); Shen Zhen Wingor Biotechnology CO. LTD (Industry)
Responsible Party: Principal Investigator, Shi Ming, Department of Infectious Diseases, Fifth Medical Center of Chinese PLA General Hospital, National Clinical Research Center for Infectious Diseases, Beijing 302 Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022YFC2304402
Record Dates: First submitted 2023-07-24; First posted 2023-08-14 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Acute-On-Chronic Liver Failure
Keywords: Mesenchymal Stem Cells; Acute-On-Chronic Liver Failure; Therapeutics
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Control (Placebo Comparator): standard medical treatment+Placebo(5% human serum albumin in 0.9% saline, at week0, week1 and week2)
  Interventions: Drug: standard medical treatment; Drug: Placebo
- Group MSC-1 (Experimental): Patients received standard medical treatment and infusions of hUC-MSC(1.5×10^8) via peripheral veins once a week for 3 timess(at week0, week1, and week2).
  Interventions: Drug: standard medical treatment; Drug: hUC-MSC
- Group MSC-2 (Experimental): Patients in Group MSC-1 received standard medical treatment and infusions of hUC-MSC(1.5×10^8) via peripheral veins once a week for another 2 timess(at week4 and week5).
  Interventions: Drug: standard medical treatment; Drug: hUC-MSC; Drug: hUC-MSC_Prolonged

INTERVENTIONS:
Drug: standard medical treatment — standard medical treatment for ACLF
Drug: Placebo — 5% human serum albumin in 0.9% saline (at week0, week1 and week2)
  Arms: Group Control
Drug: hUC-MSC — hUC-MSC (1.5×10^8 cells/time, Peripheral IV, at week0, week1 and week2)
  Arms: Group MSC-1; Group MSC-2
Drug: hUC-MSC_Prolonged — hUC-MSC (1.5×10^8 cells/time, Peripheral IV, at week4 and week5)
  Arms: Group MSC-2

SUMMARY:
This study is a randomized double-blind placebo-controlled multicenter clinical trial to evaluate the safety and efficacy of human umbilical cord mesenchymal stem cell (UC-MSC) transplantation for the treatment of acute-on-chronic liver failure (ACLF). UC-MSC therapy may improve the clinical outcomes of patients with ACLF. The trial would provide scientific evidence for UC-MSC transplantation as a potential treatment for ACLF.

DETAILED DESCRIPTION:
Acute-on-chronic liver failure (ACLF) has been proposed to define a distinct syndrome which is characterized by an intense systemic inflammatory response, single- or multiple organ system failures, and high 28-day mortality. Current treatments for liver failure are still limited, and liver transplantation remains the only available approach to improve survival but is restricted by a shortage of organ resources, rejection after transplantation, and heavy financial costs. In the past decade, a series of new applications based on mesenchymal stem cell (MSC) therapy have been studied as an alternative interventional method for chronic liver diseases. This randomized double-blind placebo-controlled multicenter clinical trial is aimed at determining the safety and clinical efficacy of UC-MSC transfusions in ACLF patients.

A total of 150 ACLF patients would be enrolled,100patients would be assigned to the MSC intervention group and the other 50 patients would be assigned to the placebo control group. This trial is two-stage randomized designed. At the first stage, the patients would be randomized into two groups, the placebo short control group would receive standard medical treatment plus 3 times placebo (at week0, week1 and week2), while the MSC short treatment group would receive standard medical treatment plus 3 times hUC-MSC (1.5×10^8, Peripheral IV, at week0, week1 and week2). The two groups would be followed up for 2 weeks, and unblinding would be conducted at week4. At the second stage, the survived patients of the MSC short treatment group would be further randomized and blinded into another two groups. The MSC Prolonged treatment group would receive another 2 times hUC-MSC (1.5×10^8, Peripheral IV, at week4 and week5), while the MSC Prolonged control group would receive 2 times placebo (at week4 and week5).

Transplantation free survival rate and incidence of treatment-emergent adverse events would be the primary outcomes, and other outcomes such as international normalized ratio (INR), total bilirubin (TBIL, mg/dL), serum albumin (ALB, g/L), blood urea nitrogen (BUN, mmol/l), the model for end-stage liver disease(MELD) score and child-turcotte-pugh(CTP) score would also be measured.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old ≤ age ≤ 70 years old, gender is not limited.
2. Meet the APASL definition of ACLF: acute liver injury in patients with previously diagnosed or undiagnosed chronic liver disease or cirrhosis, manifested as jaundice (total bilirubin levels of 5 mg/dl or more) and coagulopathy (INR of 1.5 or more, or prothrombin activity of less than 40%） complicated within 4 weeks by clinical ascites, encephalopathy, or both.
3. Willing to sign the informed consent form.

Exclusion Criteria:

1. Patients with acute kidney injury, upper gastrointestinal hemorrhage, hepatic encephalopathy above grade II (inclusive) or uncontrolled infection at baseline;
2. Before the onset of liver failure, the previous indicators of the patient included PLT<50×10^9/L or Child-Pugh score>9;
3. Combined with liver cancer or other malignant tumors;
4. Patients with previous liver transplantation or planned liver transplantation within 3 months;
5. Severe organic disease of primary extrahepatic organs;
6. Those who have a history of venous thrombosis or pulmonary embolism are judged by the investigator to be ineligible to participate in this trial;
7. Pregnant, breastfeeding women or those who plan to have a baby in the near future;
8. Those who are highly allergic or have a history of severe allergies;
9. Those who have received immunosuppressant and immune enhancer treatment within 1 month;
10. Drug abuse in the past 5 years;
11. Alcohol withdrawal symptoms;
12. A history of severe mental disorders within 24 months before screening, including uncontrolled major depression or controlled or uncontrolled psychosis;
13. Those who have participated or are participating in other clinical trials within three months before screening, or have previously received stem cell therapy;
14. Other conditions that the investigator thinks that the patient is not suitable to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Transplantation free survival rate | week1, week2, week3, week4, week5, week8, week12, week24, week53
  Transplantation free survival rate of ACLF patients.
Incidence of Treatment-Emergent Adverse Events | day0, day3, week1, week2, week3, week4, week5, week8, week12, week24, week53
  Safety and Tolerability of UC-MSCs transplantation.

SECONDARY OUTCOMES:
International Normalized Ratio (INR) | week-1, week0, day3, week1, week2, week3, week4, week5, week12, week24, week53
  INR was introduced as a standardized reporting mechanism allowing comparisons across laboratories and patients. Consensus guidelines recommend that INR ≥ 1.5 can be used as a threshold, and current recommendations for targeting an INR of < 1.5 were based on studies across all surgical disciplines.
Concentration of Total Bilirubin (TBIL, mg/dL) | week-1, week0, day3, week1, week2, week3, week4, week5, week12, week24, week53
  Total bilirubin refers to the concentration of bilirubin in a patient's blood sample, which is automatically measured by the laboratories in accordance with standard operating procedures. APASL defines ACLF as "an acute hepatic insult manifesting as jaundice (Serum Bilirubin ≥ 5 mg/dL) and coagulopathy (international normalized ratio [INR] ≥ 1.5) complicated within 4 weeks by clinical ascites and/or encephalopathy in a patient with previously diagnosed or undiagnosed chronic liver disease/cirrhosis, that is associated with a high 28-day mortality."
Concentration of Serum Albumin (ALB, g/L) | week-1, week0, day3, week1, week2, week3, week4, week5, week12, week24, week53
  Serum albumin refers to the concentration of albumin in a patient's serum, which is automatically measured by the laboratory in accordance with standard operating procedures. Serum albumin is an independent protective factor for 30-day prognosis in ACLF patients.
Concentration of Blood Urea Nitrogen (BUN, mmol/L) | week-1, week0, day3, week1, week2, week3, week4, week5, week12, week24, week53
  Blood urea nitrogen refers to the concentration of urea nitrogen in a patient's blood sample. Blood urea nitrogen is a commonly used indicator of renal function in clinic.
The Model for End-Stage Liver Disease(MELD) score | week-1, week1, week2, week4, week5, week12, week24, week53
  R = 3.8×ln [TBiL (mg/dl)] +11.2×ln (INR) +9.6×ln [Cr (mg/dl)] +6.4× (Cause: biliary or alcoholic is 0, other is 1), the result is taken as an integer. Studies have shown that the optimal critical value of MELD score to judge the short-term prognosis of ACLF patients is 30, and when MELD score is greater than 30, the case fatality rate of patients within 3 months is significantly increased.
Child-Turcotte-Pugh(CTP) score | week-1, week1, week2, week4, week5, week12, week24, week53
  CTP score is currently the most commonly used model to evaluate liver reserve function and prognosis in patients with cirrhosis. This model evaluates liver function based on HE grade, degree of abdominal fluid accumulation, bilirubin (TBiL), albumin (Alb) and prothrombin time (PT). The score ranges from 0 to 15, with the higher the score, the worse the prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, PhD, Principal Investigator — the Fifth Medical Center, Chinese PLA General Hospital
Locations (1):
- the Fifth Medical Center, Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin BL, Chen JF, Qiu WH, Wang KW, Xie DY, Chen XY, Liu QL, Peng L, Li JG, Mei YY, Weng WZ, Peng YW, Cao HJ, Xie JQ, Xie SB, Xiang AP, Gao ZL. Allogeneic bone marrow-derived mesenchymal stromal cells for hepatitis B virus-related acute-on-chronic liver failure: A randomized controlled trial. Hepatology. 2017 Jul;66(1):209-219. doi: 10.1002/hep.29189. Epub 2017 May 27. PMID 28370357
- [Background] Schacher FC, Martins Pezzi da Silva A, Silla LMDR, Alvares-da-Silva MR. Bone Marrow Mesenchymal Stem Cells in Acute-on-Chronic Liver Failure Grades 2 and 3: A Phase I-II Randomized Clinical Trial. Can J Gastroenterol Hepatol. 2021 Aug 4;2021:3662776. doi: 10.1155/2021/3662776. eCollection 2021. PMID 34395335
- [Background] Xu WX, He HL, Pan SW, Chen YL, Zhang ML, Zhu S, Gao ZL, Peng L, Li JG. Combination Treatments of Plasma Exchange and Umbilical Cord-Derived Mesenchymal Stem Cell Transplantation for Patients with Hepatitis B Virus-Related Acute-on-Chronic Liver Failure: A Clinical Trial in China. Stem Cells Int. 2019 Feb 4;2019:4130757. doi: 10.1155/2019/4130757. eCollection 2019. PMID 30863450
- [Background] Shi M, Zhang Z, Xu R, Lin H, Fu J, Zou Z, Zhang A, Shi J, Chen L, Lv S, He W, Geng H, Jin L, Liu Z, Wang FS. Human mesenchymal stem cell transfusion is safe and improves liver function in acute-on-chronic liver failure patients. Stem Cells Transl Med. 2012 Oct;1(10):725-31. doi: 10.5966/sctm.2012-0034. Epub 2012 Oct 11. PMID 23197664
- [Background] Li YH, Xu Y, Wu HM, Yang J, Yang LH, Yue-Meng W. Umbilical Cord-Derived Mesenchymal Stem Cell Transplantation in Hepatitis B Virus Related Acute-on-Chronic Liver Failure Treated with Plasma Exchange and Entecavir: a 24-Month Prospective Study. Stem Cell Rev Rep. 2016 Dec;12(6):645-653. doi: 10.1007/s12015-016-9683-3. PMID 27687792
- [Background] Yu H, Feng Y, Du W, Zhao M, Jia H, Wei Z, Yan S, Han Z, Zhang L, Li Z, Han Z. Off-the-shelf GMP-grade UC-MSCs as therapeutic drugs for the amelioration of CCl4-induced acute-on-chronic liver failure in NOD-SCID mice. Int Immunopharmacol. 2022 Dec;113(Pt A):109408. doi: 10.1016/j.intimp.2022.109408. Epub 2022 Nov 9. PMID 36461584
- [Background] Gilsanz C, Aller MA, Fuentes-Julian S, Prieto I, Blazquez-Martinez A, Argudo S, Fernandez-Delgado J, Belena J, Arias J, De Miguel MP. Adipose-derived mesenchymal stem cells slow disease progression of acute-on-chronic liver failure. Biomed Pharmacother. 2017 Jul;91:776-787. doi: 10.1016/j.biopha.2017.04.117. Epub 2017 May 10. PMID 28501004
- [Background] Maheshwari D, Kumar D, Jagdish RK, Nautiyal N, Hidam A, Kumari R, Sehgal R, Trehanpati N, Baweja S, Kumar G, Sinha S, Bajpai M, Pamecha V, Bihari C, Maiwall R, Sarin SK, Kumar A. Bioenergetic Failure Drives Functional Exhaustion of Monocytes in Acute-on-Chronic Liver Failure. Front Immunol. 2022 Jun 3;13:856587. doi: 10.3389/fimmu.2022.856587. eCollection 2022. PMID 35747140
- [Background] He Y, Guo X, Lan T, Xia J, Wang J, Li B, Peng C, Chen Y, Hu X, Meng Z. Human umbilical cord-derived mesenchymal stem cells improve the function of liver in rats with acute-on-chronic liver failure via downregulating Notch and Stat1/Stat3 signaling. Stem Cell Res Ther. 2021 Jul 13;12(1):396. doi: 10.1186/s13287-021-02468-6. PMID 34256837
- [Background] Lin D, Chen H, Xiong J, Zhang J, Hu Z, Gao J, Gao B, Zhang S, Chen J, Cao H, Li Z, Lin B, Gao Z. Mesenchymal stem cells exosomal let-7a-5p improve autophagic flux and alleviate liver injury in acute-on-chronic liver failure by promoting nuclear expression of TFEB. Cell Death Dis. 2022 Oct 12;13(10):865. doi: 10.1038/s41419-022-05303-9. PMID 36224178
- [Derived] Wang Y, Li M, Yang T, Xie Y, Wang FS, Hu J, Shi M. Human umbilical cord mesenchymal stem cell transplantation for the treatment of acute-on-chronic liver failure: protocol for a multicentre random double-blind placebo-controlled trial. BMJ Open. 2024 Jun 25;14(6):e084237. doi: 10.1136/bmjopen-2024-084237. PMID 38925694